CLINICAL TRIAL: NCT02765750
Title: Study of the Effect of Intraoperative Positive Messages on Postoperative Outcomes
Brief Title: Postoperative Outcomes After Positive Intraoperative Messages
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary investigator was transferred to another hospital
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Georgios Kotsovolis, Dr, 424 General Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4659
Record Dates: First submitted 2016-04-29; First posted 2016-05-09 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain; Postoperative Nausea; Postoperative Vomiting
Keywords: Emergence agitation
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Emergence Delirium | interventions — NMT1 protein, S pombe

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIS 40-60 (Experimental): Patient with intraoperative Bispectral Index (BIS) 40-60.
  Interventions: Behavioral: Intraoperative positive messages
- BIS 20-40 (Experimental): Patient with intraoperative Bispectral Index (BIS) 20-40.
  Interventions: Behavioral: Intraoperative positive messages
- Placebo (Placebo Comparator): Placebo group
  Interventions: Behavioral: No message

INTERVENTIONS:
Behavioral: Intraoperative positive messages — The message "You are in the operating room. Everything is going very well. When you wake up you will be very calm, you will not feel pain and you will not have nausea" will be played in greek language by headphones to the patient when the Bispectral Index (BIS) is 40-60.
  Arms: BIS 40-60
Behavioral: Intraoperative positive messages — The message "You are in the operating room. Everything is going very well. When you wake up you will be very calm, you will not feel pain and you will not have nausea" will be played in greek language by headphones to the patient when the Bispectral Index (BIS) is 20-40.
  Arms: BIS 20-40
Behavioral: No message — The headphones will be placed on patient's ears but no message will be played.
  Arms: Placebo

SUMMARY:
The patients scheduled for laparoscopic cholecystectomy will be allocated to 3 groups. Group A and B patients will listen to a positive message under general anesthesia. Group C patients will not listen to the message. The postoperative pain, analgesic consumption and frequency of nausea, vomiting and emergence agitation episodes will be documented and compared between the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy.
* ASA 1-3

Exclusion Criteria:

* Hearing loss.
* Chronic use of drugs which affect the central nervous system (antidepressants, antiepileptics, opioids, benzodiazepines)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03; Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity. | Within an average of 15 minutes after emergence from general anesthesia.
  The patients will be asked to evaluate their postoperative pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain). Pain will be evaluated in supine position, after cough and after change of position from supine to standing.
Postoperative paracetamol consumption. | 24 hours after emergence from general anesthesia.
  The patients will be instructed to ask for analgesics as needed. When rescue analgesia is required 1000mg paracetamol will be administered. The frequency of paracetamol administration will be documented.
Postoperative tramadol consumption. | 24 hours after emergence from general anesthesia.
  If the administration of paracetamol doesn't relieve postoperative pain and the patients continues to ask for analgesia, 100mg tramadol will be administered. The frequency of tramadol administration will be documented.
Emergence agitation (yes/no). | Within an average of 10 minutes after emergence from general anesthesia.
  The patients' mental status will be evaluated with the 7grade Riker's Agitation-Sedation Scale. If the patient has a score of 5 or greater he will be documented as a case of emergence agitation.
Postoperative nausea. | 24 hours after emergence from general anesthesia.
  The frequency of episodes of nausea will be documented.
Postoperative vomiting. | 24 hours after emergence from general anesthesia.
  The frequency of episodes of vomiting will be documented.
Pain Intensity. | 1 hour after the end of surgery.
  The patients will be asked to evaluate their postoperative pain by using the 11 grade Numerical Rating Scale (0 no pain, 10 maximum possible pain). Pain will be evaluated in supine position, after cough and after change of position from supine to standing.
Pain Intensity. | 6 hours after the end of surgery.
  Numerical Rating Scale (0 no pain, 10 maximum possible pain). Pain will be evaluated in supine position, after cough and after change of position from supine to standing.
Pain Intensity. | 12 hours after the end of surgery.
  Numerical Rating Scale (0 no pain, 10 maximum possible pain). Pain will be evaluated in supine position, after cough and after change of position from supine to standing.
Pain Intensity. | 24 hours after the end of surgery.
  Numerical Rating Scale (0 no pain, 10 maximum possible pain). Pain will be evaluated in supine position, after cough and after change of position from supine to standing.

SECONDARY OUTCOMES:
Explicit memory. | 24 hours after emergence from general anesthesia.
  The patient will be asked to answer the modified Brice questionnaire in order to investigate for explicit memory of the intraoperative message or other events.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Kotsovolis, Dr, Principal Investigator — 424 Army General Hospital
Locations (1):
- 424 Army General Hospital Department of Anesthesia, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdeshahi SK, Hashemipour MA, Mesgarzadeh V, Shahidi Payam A, Halaj Monfared A. Effect of hypnosis on induction of local anaesthesia, pain perception, control of haemorrhage and anxiety during extraction of third molars: a case-control study. J Craniomaxillofac Surg. 2013 Jun;41(4):310-5. doi: 10.1016/j.jcms.2012.10.009. Epub 2012 Dec 14. PMID 23253486
- [Background] Aberg KC, Albrecht E, Tartaglia EM, Farron A, Soom P, Herzog MH. Anesthesia prevents auditory perceptual learning. Anesthesiology. 2009 Nov;111(5):1010-5. doi: 10.1097/01.anes.0000363310.19041.90. PMID 19858871
- [Background] Aceto P, Valente A, Gorgoglione M, Adducci E, De Cosmo G. Relationship between awareness and middle latency auditory evoked responses during surgical anaesthesia. Br J Anaesth. 2003 May;90(5):630-5. doi: 10.1093/bja/aeg113. PMID 12697591
- [Background] Aceto P, Lai C, Perilli V, Dello Russo C, Federico B, Navarra P, Proietti R, Sollazzi L. Stress-related biomarkers of dream recall and implicit memory under anaesthesia. Anaesthesia. 2013 Nov;68(11):1141-7. doi: 10.1111/anae.12386. Epub 2013 Aug 19. PMID 23952901
- [Background] Andrade J. Does memory priming during anesthesia matter? Anesthesiology. 2005 Nov;103(5):919-20. doi: 10.1097/00000542-200511000-00002. No abstract available. PMID 16249662
- [Background] Andrade J. Investigations of hypesthesia: using anesthetics to explore relationships between consciousness, learning, and memory. Conscious Cogn. 1996 Dec;5(4):562-80. doi: 10.1006/ccog.1996.0033. PMID 9063616
- [Background] Andrade J. Learning during anaesthesia: a review. Br J Psychol. 1995 Nov;86 ( Pt 4):479-506. doi: 10.1111/j.2044-8295.1995.tb02566.x. PMID 8542198
- [Background] Andrade J, Deeprose C. Unconscious memory formation during anaesthesia. Best Pract Res Clin Anaesthesiol. 2007 Sep;21(3):385-401. doi: 10.1016/j.bpa.2007.04.006. PMID 17900016
- [Background] American Society of Anesthesiologists Task Force on Intraoperative Awareness. Practice advisory for intraoperative awareness and brain function monitoring: a report by the american society of anesthesiologists task force on intraoperative awareness. Anesthesiology. 2006 Apr;104(4):847-64. doi: 10.1097/00000542-200604000-00031. No abstract available. PMID 16571982
- [Background] Bailey AR, Jones JG. Patients' memories of events during general anaesthesia. Anaesthesia. 1997 May;52(5):460-76. doi: 10.1111/j.1365-2044.1997.133-az0134.x. PMID 9165967
- [Background] Barr G, Anderson RE, Owall A, Jakobsson JG. Being awake intermittently during propofol-induced hypnosis: a study of BIS, explicit and implicit memory. Acta Anaesthesiol Scand. 2001 Aug;45(7):834-8. doi: 10.1034/j.1399-6576.2001.045007834.x. PMID 11472283
- [Background] Bejjani G, Lequeux PY, Schmartz D, Engelman E, Barvais L. No evidence of memory processing during propofol-remifentanil target-controlled infusion anesthesia with bispectral index monitoring in cardiac surgery. J Cardiothorac Vasc Anesth. 2009 Apr;23(2):175-81. doi: 10.1053/j.jvca.2008.09.016. Epub 2008 Nov 20. PMID 19026570
- [Background] Bennett HL, Davis HS, Giannini JA. Non-verbal response to intraoperative conversation. Br J Anaesth. 1985 Feb;57(2):174-9. doi: 10.1093/bja/57.2.174. PMID 3970796
- [Background] Block RI, Ghoneim MM, Sum Ping ST, Ali MA. Efficacy of therapeutic suggestions for improved postoperative recovery presented during general anesthesia. Anesthesiology. 1991 Nov;75(5):746-55. doi: 10.1097/00000542-199111000-00005. PMID 1952199
- [Background] Block RI, Ghoneim MM, Sum Ping ST, Ali MA. Human learning during general anaesthesia and surgery. Br J Anaesth. 1991 Feb;66(2):170-8. doi: 10.1093/bja/66.2.170. PMID 1817616
- [Background] Block RI, Ghoneim MM. Insensitivity of implicit memory to anesthesia methods. Anesthesiology. 1994 Aug;81(2):516-7. doi: 10.1097/00000542-199408000-00036. No abstract available. PMID 8053605
- [Background] Boeke S, Bonke B, Bouwhuis-Hoogerwerf ML, Bovill JG, Zwaveling A. Effects of sounds presented during general anaesthesia on postoperative course. Br J Anaesth. 1988 May;60(6):697-702. doi: 10.1093/bja/60.6.697. PMID 3377953
- [Background] Bonebakker AE, Bonke B, Klein J, Wolters G, Stijnen T, Passchier J, Merikle PM. Information processing during general anesthesia: evidence for unconscious memory. Mem Cognit. 1996 Nov;24(6):766-76. doi: 10.3758/bf03201101. PMID 8961821
- [Background] Bonebakker AE, Jelicic M, Passchier J, Bonke B. Memory during general anesthesia: practical and methodological aspects. Conscious Cogn. 1996 Dec;5(4):542-61. doi: 10.1006/ccog.1996.0032. PMID 9063615
- [Background] Bonett E, Pham X, Smith KR, Howard K, Sheppard S, Davidson A. Implicit memory formation using the word stem completion task during anesthesia in children. Paediatr Anaesth. 2014 Mar;24(3):290-6. doi: 10.1111/pan.12299. Epub 2013 Nov 13. PMID 24219512
- [Background] Del Casale A, Ferracuti S, Rapinesi C, Serata D, Caltagirone SS, Savoja V, Piacentino D, Callovini G, Manfredi G, Sani G, Kotzalidis GD, Girardi P. Pain perception and hypnosis: findings from recent functional neuroimaging studies. Int J Clin Exp Hypn. 2015;63(2):144-70. doi: 10.1080/00207144.2015.1002371. PMID 25719519
- [Background] Cascella M. What about Memory, Consciousness, Recall, and Awareness in Anesthesia? Iran J Med Sci. 2014 May;39(3):311-2. No abstract available. PMID 24850992
- [Background] Cheng CM, Huang CL. Processes of conscious and unconscious memory: evidence from current research on dissociation of memories within a test. Am J Psychol. 2011 Winter;124(4):421-40. doi: 10.5406/amerjpsyc.124.4.0421. PMID 22324282
- [Background] Dawson P, Van Hamel C, Wilkinson D, Warwick P, O'Connor M. Patient-controlled analgesia and intra-operative suggestion. Anaesthesia. 2001 Jan;56(1):65-9. doi: 10.1046/j.1365-2044.2001.01763-5.x. PMID 11167439
- [Background] Deeprose C, Andrade J, Harrison D, Edwards N. Unconscious auditory priming during surgery with propofol and nitrous oxide anaesthesia: a replication. Br J Anaesth. 2005 Jan;94(1):57-62. doi: 10.1093/bja/aeh289. Epub 2004 Oct 14. PMID 15486010
- [Background] Deeprose C, Andrade J, Varma S, Edwards N. Unconscious learning during surgery with propofol anaesthesia. Br J Anaesth. 2004 Feb;92(2):171-7. doi: 10.1093/bja/aeh054. PMID 14722165
- [Background] Deeprose C, Andrade J. Is priming during anesthesia unconscious? Conscious Cogn. 2006 Mar;15(1):1-23. doi: 10.1016/j.concog.2005.05.003. Epub 2005 Jul 25. PMID 16043367
- [Background] Dobrunz UE, Jaeger K, Vetter G. Memory priming during light anaesthesia with desflurane and remifentanil anaesthesia. Br J Anaesth. 2007 Apr;98(4):491-6. doi: 10.1093/bja/aem008. Epub 2007 Feb 27. PMID 17327251
- [Background] Evans C, Richardson PH. Improved recovery and reduced postoperative stay after therapeutic suggestions during general anaesthesia. Lancet. 1988 Aug 27;2(8609):491-3. doi: 10.1016/s0140-6736(88)90131-6. PMID 2900410
- [Background] Flouda L, Pandazi A, Papageorgiou C, Perrea D, Krepi E, Kostopanagiotou G. Comparative effects of sevoflurane and propofol based general anaesthesia for elective surgery on memory. Arch Med Sci. 2013 Feb 21;9(1):105-11. doi: 10.5114/aoms.2013.33351. PMID 23515343
- [Background] Fowler SL, Rasinski HM, Geers AL, Helfer SG, France CR. Concept priming and pain: an experimental approach to understanding gender roles in sex-related pain differences. J Behav Med. 2011 Apr;34(2):139-47. doi: 10.1007/s10865-010-9291-7. Epub 2010 Sep 28. PMID 20878354
- [Background] Ghoneim MM, Block RI, Dhanaraj VJ, Todd MM, Choi WW, Brown CK. Auditory evoked responses and learning and awareness during general anesthesia. Acta Anaesthesiol Scand. 2000 Feb;44(2):133-43. doi: 10.1034/j.1399-6576.2000.440202.x. PMID 10695905
- [Background] Ghoneim MM. Drugs and human memory (part 1): Clinical, theoretical, and methodologic issues. Anesthesiology. 2004 Apr;100(4):987-1002. doi: 10.1097/00000542-200404000-00033. No abstract available. PMID 15087638
- [Background] Ghoneim MM, Block RI. Learning and memory during general anesthesia: an update. Anesthesiology. 1997 Aug;87(2):387-410. doi: 10.1097/00000542-199708000-00027. No abstract available. PMID 9286904
- [Background] Goldmann L, Shah MV, Hebden MW. Memory of cardiac anaesthesia. Psychological sequelae in cardiac patients of intra-operative suggestion and operating room conversation. Anaesthesia. 1987 Jun;42(6):596-603. doi: 10.1111/j.1365-2044.1987.tb03082.x. PMID 3618993
- [Background] Hadzidiakos D, Horn N, Degener R, Buchner A, Rehberg B. Analysis of Memory Formation during General Anesthesia (Propofol/Remifentanil) for Elective Surgery Using the Process-dissociation Procedure. Anesthesiology. 2009 Aug;111(2):293-301. doi: 10.1097/ALN.0b013e3181ac4a4b. PMID 19568158
- [Background] Hughes JA, Sanders LD, Dunne JA, Tarpey J, Vickers MD. Reducing smoking. The effect of suggestion during general anaesthesia on postoperative smoking habits. Anaesthesia. 1994 Feb;49(2):126-8. doi: 10.1111/j.1365-2044.1994.tb03368.x. PMID 7864913
- [Background] Iselin-Chaves IA, Willems SJ, Jermann FC, Forster A, Adam SR, Van der Linden M. Investigation of implicit memory during isoflurane anesthesia for elective surgery using the process dissociation procedure. Anesthesiology. 2005 Nov;103(5):925-33. doi: 10.1097/00000542-200511000-00005. PMID 16249665
- [Background] Jelicic M, Bonke B. Implicit memory for stimuli presented during anaesthesia: role of anaesthetic cocktail and memory test. Med Hypotheses. 1993 Oct;41(4):353-4. doi: 10.1016/0306-9877(93)90082-2. PMID 8289702
- [Background] Jelicic M, Bonke B, Millar K. Effect of different therapeutic suggestions presented during anaesthesia on post-operative course. Eur J Anaesthesiol. 1993 Sep;10(5):343-7. PMID 11767423
- [Background] Kekecs Z, Nagy T, Varga K. The effectiveness of suggestive techniques in reducing postoperative side effects: a meta-analysis of randomized controlled trials. Anesth Analg. 2014 Dec;119(6):1407-19. doi: 10.1213/ANE.0000000000000466. PMID 25289661
- [Background] Kendrick C, Sliwinski J, Yu Y, Johnson A, Fisher W, Kekecs Z, Elkins G. Hypnosis for Acute Procedural Pain: A Critical Review. Int J Clin Exp Hypn. 2016;64(1):75-115. doi: 10.1080/00207144.2015.1099405. PMID 26599994
- [Background] Kerssens C, Klein J, van der Woerd A, Bonke B. Auditory information processing during adequate propofol anesthesia monitored by electroencephalogram bispectral index. Anesth Analg. 2001 May;92(5):1210-4. doi: 10.1097/00000539-200105000-00024. PMID 11323348
- [Background] Kerssens C. Implicit memory phenomena under anesthesia are not spurious. Anesthesiology. 2010 Mar;112(3):764-5; author reply 765-6. doi: 10.1097/ALN.0b013e3181cf3ffc. No abstract available. PMID 20179526
- [Background] Kerssens C, Lubke GH, Klein J, van der Woerd A, Bonke B. Memory function during propofol and alfentanil anesthesia: predictive value of individual differences. Anesthesiology. 2002 Aug;97(2):382-9. doi: 10.1097/00000542-200208000-00015. PMID 12151928
- [Background] Kerssens C. Using the process dissociation procedure: the meaning and value of comparable base rates. Anesthesiology. 2007 Jul;107(1):172-3; author reply 174. doi: 10.1097/01.anes.0000268505.82823.f3. No abstract available. PMID 17585238
- [Background] Kerssens C, Gaither JR, Sebel PS. Preserved memory function during bispectral index-guided anesthesia with sevoflurane for major orthopedic surgery. Anesthesiology. 2009 Sep;111(3):518-24. doi: 10.1097/ALN.0b013e3181b05f0b. PMID 19672180
- [Background] Kerssens C, Ouchi T, Sebel PS. No evidence of memory function during anesthesia with propofol or isoflurane with close control of hypnotic state. Anesthesiology. 2005 Jan;102(1):57-62. doi: 10.1097/00000542-200501000-00012. PMID 15618787
- [Background] Kessels RP, Remmerswaal M, Wilson BA. Assessment of nondeclarative learning in severe Alzheimer dementia: the Implicit Memory Test (IMT). Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):179-83. doi: 10.1097/WAD.0b013e318203f3ab. PMID 21192238
- [Background] Kurata J, Hemmings HC Jr. Memory and awareness in anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i1-i3. doi: 10.1093/bja/aev224. No abstract available. PMID 26174293
- [Background] van der Laan WH, van Leeuwen BL, Sebel PS, Winograd E, Baumann P, Bonke B. Therapeutic suggestion has not effect on postoperative morphine requirements. Anesth Analg. 1996 Jan;82(1):148-52. doi: 10.1097/00000539-199601000-00027. PMID 8712392
- [Background] Lebovits AH, Twersky R, McEwan B. Intraoperative therapeutic suggestions in day-case surgery: are there benefits for postoperative outcome? Br J Anaesth. 1999 Jun;82(6):861-6. doi: 10.1093/bja/82.6.861. PMID 10562780
- [Background] Leclerc C, Gerard JL, Bricard H. [Intraoperative memory. A study of its incidence in general anesthesia in 326 patients]. Ann Fr Anesth Reanim. 2001 Aug;20(7):592-9. doi: 10.1016/s0750-7658(01)00446-4. French. PMID 11530746
- [Background] Lequeux PY, Bejjani G, Sekkat H. Implicit memory during isoflurane anesthesia. Anesthesiology. 2006 Aug;105(2):429; author reply 430. doi: 10.1097/00000542-200608000-00032. No abstract available. PMID 16871083
- [Background] Lequeux PY, Hecquet F, Bredas P. Does anesthetic regimen influence implicit memory during general anesthesia? Anesth Analg. 2014 Nov;119(5):1174-9. doi: 10.1213/ANE.0000000000000162. PMID 24797121
- [Background] Liu WH, Standen PJ, Aitkenhead AR. Therapeutic suggestions during general anaesthesia in patients undergoing hysterectomy. Br J Anaesth. 1992 Mar;68(3):277-81. doi: 10.1093/bja/68.3.277. PMID 1547052
- [Background] Lubke GH, Kerssens C, Phaf H, Sebel PS. Dependence of explicit and implicit memory on hypnotic state in trauma patients. Anesthesiology. 1999 Mar;90(3):670-80. doi: 10.1097/00000542-199903000-00007. PMID 10078666
- [Background] Lubke GH, Kerssens C, Gershon RY, Sebel PS. Memory formation during general anesthesia for emergency cesarean sections. Anesthesiology. 2000 Apr;92(4):1029-34. doi: 10.1097/00000542-200004000-00020. PMID 10754622
- [Background] Lubke GH, Sebel PS. Awareness and different forms of memory in trauma anaesthesia. Curr Opin Anaesthesiol. 2000 Apr;13(2):161-5. doi: 10.1097/00001503-200004000-00013. PMID 17016296
- [Background] Mashour GA, Avidan MS. Intraoperative awareness: controversies and non-controversies. Br J Anaesth. 2015 Jul;115 Suppl 1:i20-i26. doi: 10.1093/bja/aev034. Epub 2015 Mar 3. PMID 25735710
- [Background] McLintock TT, Aitken H, Downie CF, Kenny GN. Postoperative analgesic requirements in patients exposed to positive intraoperative suggestions. BMJ. 1990 Oct 6;301(6755):788-90. doi: 10.1136/bmj.301.6755.788. PMID 2224266
- [Background] Millar K. Efficacy of therapeutic suggestions presented during anaesthesia: re-analysis of conflicting results. Br J Anaesth. 1993 Oct;71(4):597-601. doi: 10.1093/bja/71.4.597. PMID 8260315
- [Background] Munte S, Schmidt M, Meyer M, Nager W, Lullwitz E, Munte TF, Piepenbrock S. Implicit memory for words played during isoflurane- or propofol-based anesthesia: the lexical decision task. Anesthesiology. 2002 Mar;96(3):588-94. doi: 10.1097/00000542-200203000-00013. PMID 11873032
- [Background] Munte S, Kobbe I, Demertzis A, Lullwitz E, Munte TF, Piepenbrock S, Leuwer M. Increased reading speed for stories presented during general anesthesia. Anesthesiology. 1999 Mar;90(3):662-9. doi: 10.1097/00000542-199903000-00006. PMID 10078665
- [Background] Munte S, Lullwitz E, Leuwer M, Mitzlaff B, Munte TF, Hussein S, Piepenbrock SA. No implicit memory for stories played during isoflurane/alfentanil/nitrous oxide anesthesia: a reading speed measurement. Anesth Analg. 2000 Mar;90(3):733-8. doi: 10.1097/00000539-200003000-00041. PMID 10702466
- [Background] Munte S, Munte TF, Mitzlaff B, Walz R, Leuwer M, Piepenbrock S. Postoperative reading speed does not indicate implicit memory in elderly cardiac patients after propofol and remifentanyl anaesthesia. Acta Anaesthesiol Scand. 2001 Jul;45(6):750-5. doi: 10.1034/j.1399-6576.2001.045006750.x. PMID 11421835
- [Background] Myles PS, Hendrata M, Layher Y, Williams NJ, Hall JL, Moloney JT, Powell J. Double-blind, randomized trial of cessation of smoking after audiotape suggestion during anaesthesia. Br J Anaesth. 1996 May;76(5):694-8. doi: 10.1093/bja/76.5.694. PMID 8688271
- [Background] Nilsson U, Rawal N, Unestahl LE, Zetterberg C, Unosson M. Improved recovery after music and therapeutic suggestions during general anaesthesia: a double-blind randomised controlled trial. Acta Anaesthesiol Scand. 2001 Aug;45(7):812-7. doi: 10.1034/j.1399-6576.2001.045007812.x. PMID 11472279
- [Background] Oddby-Muhrbeck E, Jakobsson J, Enquist B. Implicit processing and therapeutic suggestion during balanced anaesthesia. Acta Anaesthesiol Scand. 1995 Apr;39(3):333-7. doi: 10.1111/j.1399-6576.1995.tb04072.x. PMID 7793211
- [Background] Pham X, Smith KR, Sheppard SJ, Bradshaw C, Lo E, Davidson AJ. Implicit memory formation during routine anesthesia in children: a double-masked randomized controlled trial. Anesthesiology. 2010 May;112(5):1097-104. doi: 10.1097/ALN.0b013e3181d692c2. PMID 20354436
- [Background] Rauchs G, Desgranges B, Foret J, Eustache F. The relationships between memory systems and sleep stages. J Sleep Res. 2005 Jun;14(2):123-40. doi: 10.1111/j.1365-2869.2005.00450.x. PMID 15910510
- [Background] Reasor JD, Poe GR. Learning and memory during sleep and anesthesia. Int Anesthesiol Clin. 2008 Summer;46(3):105-29. doi: 10.1097/AIA.0b013e318181e513. No abstract available. PMID 18617820
- [Background] Renna M, Lang EM, Lockwood GG. The effect of sevoflurane on implicit memory: a double-blind, randomised study. Anaesthesia. 2000 Jul;55(7):634-40. doi: 10.1046/j.1365-2044.2000.01326.x. PMID 10919417
- [Background] Richter M, Schroeter C, Puensch T, Straube T, Hecht H, Ritter A, Miltner WH, Weiss T. Pain-related and negative semantic priming enhances perceived pain intensity. Pain Res Manag. 2014 Mar-Apr;19(2):69-74. doi: 10.1155/2014/425321. PMID 24716197
- [Background] Rundshagen I, Schnabel K, Schulte am Esch J. Recovery of memory after general anaesthesia: clinical findings and somatosensory evoked responses. Br J Anaesth. 2002 Mar;88(3):362-8. doi: 10.1093/bja/88.3.362. PMID 11990267
- [Background] Russell IF, Wang M. Absence of memory for intra-operative information during surgery with total intravenous anaesthesia. Br J Anaesth. 2001 Feb;86(2):196-202. doi: 10.1093/bja/86.2.196. PMID 11573659
- [Background] Sebel PS. Memory during anesthesia: gone but not forgotten? Anesth Analg. 1995 Oct;81(4):668-70. doi: 10.1097/00000539-199510000-00002. No abstract available. PMID 7573991
- [Background] Stonell CA, Leslie K, He C, Lee L. No sex differences in memory formation during general anesthesia. Anesthesiology. 2006 Nov;105(5):920-6. doi: 10.1097/00000542-200611000-00012. PMID 17065885
- [Background] Veselis RA. Gone but not forgotten-or was it? Br J Anaesth. 2004 Feb;92(2):161-3. doi: 10.1093/bja/aeh030. No abstract available. PMID 14722162
- [Background] Veselis RA. Memory formation during anaesthesia: plausibility of a neurophysiological basis. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i13-i19. doi: 10.1093/bja/aev035. Epub 2015 Mar 3. PMID 25735711
- [Background] Veselis RA. Memory function during anesthesia. Anesthesiology. 1999 Mar;90(3):648-50. doi: 10.1097/00000542-199903000-00003. No abstract available. PMID 10078662
- [Background] Veselis RA. Memory: a guide for anaesthetists. Best Pract Res Clin Anaesthesiol. 2007 Sep;21(3):297-312. doi: 10.1016/j.bpa.2007.04.002. PMID 17900010